CLINICAL TRIAL: NCT00491491
Title: SPINOZA / שפינוזה. Study With Preparatory INduction Of Zevalin in Aggressive Lymphoma. A Randomized Phase 3 Study of BEAM Versus 90Yttrium Ibritumomab Tiuxetan (Zevalin) / BEAM in Patients Requiring Autologous Hematopoietic Stem Cell Transplantation (ASCT) for Relapsed Diffuse Large B-cell Lymphoma
Brief Title: Zevalin-beam for Aggressive Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: City of Hope Medical Center (Other); Amsterdam UMC, location VUmc (Other); University of Göttingen (Other)
Responsible Party: Principal Investigator, Dr. Avichai Shimoni MD, Dr. Avichai Shimoni, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-07-4466-AN-CTIL
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: non-Hodgkin's lymphoma; autologous stem cell transplantation; radioimmunotherapy; zevalin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Z-BEAM (Experimental): ibritumomab tiuxetan (zevalin) BEAM
  Interventions: Drug: ibritumomab tiuxetan; Procedure: BEAM chemotherapy and autologous stem-cell transplantation
- standard BEAM (Active Comparator): standard BEAM chemotherapy
  Interventions: Procedure: BEAM chemotherapy and autologous stem-cell transplantation

INTERVENTIONS:
Drug: ibritumomab tiuxetan — 0.4 mCi/kg
  Other Names: zevalin
  Arms: Z-BEAM
Procedure: BEAM chemotherapy and autologous stem-cell transplantation

SUMMARY:
The study hypothesis is that the addition of zevalin radioimmunotherapy to the conditioning regimen given prior to BEAM high-dose chemotherapy and autologous stem cell transplantation in patients with aggressive lymphoma will reduced disease recurrence rate and improve overall and disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD20 positive diffuse large B-cell lymphoma as confirmed by a pathological biopsy report.
2. Patients who are candidates for autologous stem-cell transplantation due to primary refractory or first relapse of disease.
3. Patients must have chemo-sensitive disease achieving at least partial response (Cheson 2007 criteria) to last chemotherapy.
4. Age ≥ 18 years and age ≤ 70
5. Patients with adequate autologous stem cell collection for transplantation (target ≥ 2.5 x 106 CD34+ cells/kg).
6. Patients must sign written informed consent.
7. Adequate birth control in fertile patients.
8. All prior chemotherapy completed at least three weeks before study treatment.
9. Marrow involvement less than 25% at transplantation, no limitation on blood counts (low platelet count allowed).
10. Negative HIV antibody.

Exclusion Criteria:

1. 1. Chemo-refractory disease as determined by less than partial response (Cheson 2007 Criteria) to last chemotherapy.
2. Two or more relapses after initial response to induction chemotherapy.
3. High-grade transformation from earlier diagnosis of low-grade lymphoma. Patients with "De Novo" Transformed DLBCL, defined as DLBCL only on lymph node biopsy and a discordant marrow with para-trabecular small cells at first diagnosis of lymphoma, are eligible if adherent all other selection criteria.
4. Bilirubin > 3.0 mg/dl, transaminases > 3 times upper normal limit.
5. Creatinine > 2.0 mg/dl.
6. ECOG Performance status > 2.
7. Uncontrolled infection.
8. Pregnancy or lactation.
9. Abnormal lung diffusion capacity (DLCO < 40% predicted).
10. Severe cardiovascular disease; New York Heart Association (NYHA) Functional Classification ≥2.
11. Active CNS disease involvement.
12. Presence of any other malignancy or history of prior malignancy within 5 years of study entry. Within 5 years, patients treated for Stage I or II cancers are eligible provided they have a life expectancy > 5 years in relation to this prior malignance. The 5-year exclusion rule does not apply to-non melanoma skin tumors and in situ cervical cancer.
13. Pleural effusion or ascites > 1 liter.
14. Known hypersensitivity to rituximab.
15. Psychiatric conditions/disease that impair the ability to give informed consent or to adequately co-operate.
16. Prior radioimmunotherapy.
17. Prior autologous or allogeneic HSCT.
18. Active evidence of Hepatitis B or C infection; Hepatitis B surface antigen positive.
19. Patients who have had prior radiation to the lung will be excluded from the study, although mediastinal irradiation will be permitted if minimal lung is in the treatment volume.
20. Patients who have received >500cGy radiation to the kidneys will be excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avichai Shimoni, MD, Study Chair — Chaim Sheba Medical Center, Tel Hashomer, Israel; Amrita Krishnan, MD, Study Chair — City of Hope National Medical Center, Duarte, CA
Locations (9):
- United States (6):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
- Georg-August Universität, Göttingen, Germany
- Chaim Sheba Medical Center, Tel Litwinsky, Israel
- VU Medical Center, Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Z-BEAM: ibritumomab tiuxetan (zevalin) BEAM
  ibritumomab tiuxetan: 0.4 mCi/kg
  BEAM chemotherapy and autologous stem-cell transplantation
- Standard BEAM: standard BEAM chemotherapy
  BEAM chemotherapy and autologous stem-cell transplantation
Period: Overall Study
Arm/Group | Z-BEAM | Standard BEAM
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Z-BEAM | Standard BEAM | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Full Range); unit: years] | 58 [23 to 66] | 51 [24 to 67] | 55 [23 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 6 | 10 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Study stopped early due to slow accrual
  participants
    Netherlands: number analyzed (Participants) | 0 | 0 | 0
    United States: number analyzed (Participants) | 0 | 0 | 0
    Israel | 22 | 21 | 43
    Germany: number analyzed (Participants) | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: actuarial 2 year survival
Time Frame: 2 years after transplantation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Z-BEAM | Standard BEAM
Number analyzed (Participants) | 22 | 21
percentage of participants | 91 [79 to 100] | 62 [39 to 85]

2. Secondary Outcome: Progression-free Survival
Description: actuarial 2-year PFS
Time Frame: 2 years after transplantation
Measure: Number (95% Confidence Interval); unit: percentage of PARTICIPANTS
Arm/Group | Z-BEAM | Standard BEAM
Number analyzed (Participants) | 22 | 21
percentage of PARTICIPANTS | 59 [39 to 80] | 37 [14 to 60]

3. Secondary Outcome: Clinical Response
Description: complete response (CR) and partial response (PR) proportion at day 100,
Time Frame: 100 days after transplantation
Measure: Number; unit: participants
Arm/Group | Z-BEAM | Standard BEAM
Number analyzed (Participants) | 22 | 21
participants | 22 | 20

4. Secondary Outcome: Hematopoietic Recovery
Description: time to hematopoietic recovery
Time Frame: 100 days after transplantation
Measure: Median (Full Range); unit: DAYS
Arm/Group | Z-BEAM | Standard BEAM
Number analyzed (Participants) | 22 | 21
DAYS | 10 [7 to 21] | 11 [10 to 17]

5. Secondary Outcome: Grade III Toxicity
Description: incidence of infection, grade III-IV toxicities, treatment-related mortality
Time Frame: 100 days after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Z-BEAM | Standard BEAM
Number analyzed (Participants) | 22 | 21
Participants
  grade III toxicity | 3 | 4
  infection | 6 | 1
  none | 13 | 16

6. Secondary Outcome: Secondary Malignancies
Description: incidence of myelodysplastic syndrome (MDS), and secondary acute myelogenous leukemia (AML).
Time Frame: 5 years after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Z-BEAM | Standard BEAM
Number analyzed (Participants) | 22 | 21
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Z-BEAM | Standard BEAM
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/21
Other Adverse Events (participants affected / at risk) | 6/22 | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Z-BEAM (N=22) | Standard BEAM (N=21)
JC virus encephalitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Z-BEAM (N=22) | Standard BEAM (N=21)
infection (Infections and infestations) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No